CLINICAL TRIAL: NCT05939362
Title: Identifying Imaging Biomarkers Predictive of Disability Progression in Alzheimer's Disease: Pilot Study
Brief Title: New Imaging Biomarkers Predictive of MA Progression
Acronym: MR7T-PRADA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: MR7T-PRADA
Record Dates: First submitted 2023-03-01; First posted 2023-07-11 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Alzheimer Disease; Magnetic Resonance Spectroscopy; Ultra High Field 7T; Progression of Disease; MR Biomarkers
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- patient with early onset Alzheimer's disease (Experimental)
  Interventions: Other: MRI follow-up

INTERVENTIONS:
Other: MRI follow-up — MRI follow-up for patient with early onset Alzheimer's disease

SUMMARY:
The pathophysiology of AD is complex. In addition to amyloid plaques and neurofibrillary degeneration, there is a metabolic alteration of the energy pathways, oxidative phosphorylation and glycolysis, which are involved in brain function. Several authors have shown a series of early metabolic dysregulations via an increase in phosphorylation at the origin of neuronal death.

Ultra-high field imaging (7T MRI) may allow, with its better spatial resolution and advanced imaging techniques, to shed light on the mechanisms of progression of Alzheimer's disease. A Magnetic Resonance Spectroscopy (MRS) examination can be coupled to brain MRI without additional risk for the patient. Multinuclear 1H-31P metabolic imaging is a promising tool that can provide information on the metabolic evolutionary profile of AD. Thus, we propose a longitudinal study in patients with early-stage AD on 7T MRI-MRS.

ELIGIBILITY:
Inclusion Criteria:

* French-speaking patients aged 60 to 90 years,
* Patient in the context of Alzheimer's disease * for which imaging after MRI is prescribed as part of the usual diagnostic process,

  *Alzheimer's disease is diagnosed by the doctor of the memory consultation and is defined by :Evidence of a storage disorder in verbal episodic memory at LR/RI defined by a sum of LR < 17/48 and sum of RT < 40/48 +/- Impairment of executive functions possible (BREF, TMT grefex, verbal fluencies) +/- Impairment of instrumental functions possible (Grémots noun naming, Rey's figure, Mahieux's Battery).
* MMSE score ≥18,
* Written informed consent after the patient has been informed,
* Progressive decline for at least 6 months.

Exclusion Criteria:

--Partially or completely illiterate patient unable to read and write,

* Patient with an absolute contraindication to 7T MRI
* Severe psychiatric pathology not balanced,
* Non-degenerative neurological disease (stroke, multiple sclerosis ...),
* Patient with tumor or inflammatory pathology, or vascular leukopathy visualized in MRI (Fazekas score > 3)

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-10-02 (Actual); Primary Completion 2027-10-02 (Estimated); Study Completion 2028-01-15 (Estimated)

PRIMARY OUTCOMES:
To identify Magnetic Resonance Imaging biomarkers concentration (mmol/l) at baseline that are predictive of disability progression in individuals with Mild Alzheimer's disease as assessed by the Clinical Dementia Rating (CDR) scale | Baseline
  CDR scale :
  No dementia (CDR = 0), Uncertain disorders (CDR = 0.5), Mild disorders (CDR = 1), Moderate disorders (CDR = 2), Severe disorders (CDR = 3).

SECONDARY OUTCOMES:
Correlation between Imaging biomarkers concentration (mmol/l) and plasma metabolic parameters concentration (mmol/l) at baseline, Month 6 (M6) and Month 12 (M12). | up of 12 months
Correlation between Imaging biomarkers concentration (mmol/l) and Urinary metabolic parameters (mmol/l) at baseline, Month 6 (M6) and Month 12 (M12). | up of 12 months
Correlation between Imaging biomarkers concentration (mmol/l) and Enzymatic and protein parameters concentration (mmol/l) at baseline, Month 6 (M6) and Month 12 (M12). | up of 12 months
Develop realistic mathematical models that integrate multiple parameters from all generated data to predict the progression of Alzheimer's disease, as evaluated using the Clinical Dementia Rating (CDR) | up of 12 months
Build an Artificial Intelligence (AI) algorithm to predict disability progression in individuals with Mild Alzheimer's disease, as assessed by the Clinical Dementia Rating scale | up of 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Poitiers, Poitiers, France

IPD SHARING:
Plan to Share IPD: No